CLINICAL TRIAL: NCT05629871
Title: Biomarkers of Sleep-wake Cycle in Prodromal Alzheimer's Disease: Role in Cognitive Decline?
Acronym: ALZ-OREX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL18_0061
Record Dates: First submitted 2022-10-28; First posted 2022-11-29 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Neuropathology
Keywords: cognitive composite score; sleep; biomarkers; cognitive decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): Alzheimer
  Interventions: Procedure: Polysomnography; Behavioral: Neuropsychological assessment; Behavioral: Questionnaires on sleep and behavioural problems; Procedure: Actimetry; Diagnostic Test: Fractional diuresis; Procedure: Internal temperature measurement; Other: Biomarker assay

INTERVENTIONS:
Procedure: Polysomnography — Polysomnography will be performed for 24 hours at inclusion and 24 months
Behavioral: Neuropsychological assessment — A full neuropsychological assessment will be performed at inclusion, 12 and 24 months
Behavioral: Questionnaires on sleep and behavioural problems — Questionnaires on sleep and behavioural problems
Procedure: Actimetry — Measurement of actimetrics for 14 days at inclusion and at 24 months
Diagnostic Test: Fractional diuresis — Split diuresis from 7pm-7am, 7am-12am and 12pm-19pm during polysomnography at inclusion inclusion and 24 months to measure melatonin concentration
Procedure: Internal temperature measurement — eCelsius capsule to measure internal temperature at inclusion and 24 months
Other: Biomarker assay — Determination of the biomarkers Aβ42, Aβ40, Tau and P-Tau in blood and in the cerebrospinal fluid

SUMMARY:
Alzheimer's disease (AD) is characterised by a progressive loss of memory and cognitive function. In the early stages of AD, there is a progressive accumulation of molecules: β-amyloid peptides (Aβ) in the brain. There is a link between the accumulation of Aβ peptides and the deterioration of sleep, but current knowledge does not confirmed this link. The objective of this study is to define whether there is a link between cognitive decline and sleep disorders. If a correlation is found, this could allow earlier treatment of sleep disorders in the longer term in order to slow the development of AD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild Alzheimer's disease with a Mini Mental State (MMS) between 21-30
* The presence of a family carer to complete neuropsychological scales, questionnaires and sleep diaries
* Having a neurological assessment and/or follow-up requiring blood and cerebrospinal fluid (CSF) sampling with biomarkers for diagnostic purposes
* Patient who had a lumbar puncture less than one year ago or patient with a scheduled lumbar puncture as part of care
* Signed informed consent
* Able to carry out all visits and follow study procedures
* Affiliation to the French social security system

Exclusion Criteria:

* Genetic form of alzheimer's disease
* Insufficient clinical and paraclinical information for the diagnosis of AD
* Anticholinesterase and/or memantine treatment or on stable doses for at least 3 months
* Use of antidepressants, anxiolytics, hypnotics, neuroleptics, 15 days before inclusion
* Patient living in a nursing home
* Illiteracy or inability to perform psycho-behavioural tests
* Major physical or neurosensory problems that may interfere with the tests
* Initial contraindication to diagnostic lumbar puncture (LP) (spinal surgery, skin infection, haemostasis abnormality, intracranial hypertension, severe coagulation disorders, curative anticoagulant therapy, severe liver failure)
* Refusal to perform a diagnostic lumbar puncture
* Contraindication to the use of E-Celsius: people weighing less than 40 kg, with intestinal disorders, with known swallowing disorders
* Patient deprived of liberty, by judicial or administrative decision;
* Major protected by law;
* Patient in a period of relative exclusion from another protocol or for whom the maximum annual compensation of €4500 has been reached;
* Refusal to participate in the protocol.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Free and Cued Selective Reminding Test (FCSRT) scale score | From inclusion to 24 months
  The FCSRT test evaluates memory, the score obtained is between 0 and 48, higher score mean a better outcome

SECONDARY OUTCOMES:
Change in the Free and Cued Selective Reminding Test (FCSRT) scale score | From inclusion to 12 months
  The FCSRT test evaluates memory, the score obtained is between 0 and 48, higher score mean a better outcome
Cognitive decline in ADCS-PACC composite score | At inclusion and at 24 months
  The ADCS-PACC composite score is used to assess cognitive decline
Cognitive decline in the Alzheimer's Disease Cooperative Study- Preclinical Alzheimer Cognitive Composite (ADCS-PACC) composite score | At inclusion and at 12 months
  The ADCS-PACC composite score is used to assess cognitive decline
Concentration of proteins involved in Alzheimer disease | At inclusion and at 24 months
  Determination of Aβ42, Aβ40, Tau and P-Tau proteins in serum and cerebrospinal fluid
Concentration of orexinA/hypocretin | At inclusion and at 24 months
  Determination in serum and cerebrospinal fluid
Changes in sleep duration | At inclusion and at 24 months
  Average sleep duration (in hours and minutes) over a 14-day period from inclusion to M24 measured by actimetry
Sleep time at stage 1-2 during polysomnography | At inclusion and at 24 months
  Time spent in stage 1-2 sleep measured in hours and minutes during polysomnography
Sleep time at stage 3 during polysomnography | At inclusion and at 24 months
  Time spent in stage 3 sleep measured in hours and minutes during polysomnography
Time spent in Rapid eye movement (REM) sleep during polysomnography | At inclusion and at 24 months
  Time spent in stage 3 sleep measured in hours and minutes during polysomnography
Apnea Hypopnea Index | At inclusion and at 24 months
  The Apnea-Hypopnea Index is calculated from the number of apneas and hypopneas per hour of sleep (AHI = number of apneas + number of hypopneas / number of hours of sleep) during polysomnography
Nocturnal oxygen saturation (SaO2) | At inclusion and at 24 months
  The nocturnal SaO2 is an average of SaO2 values taken during the night. The value is expressed as a percentage and is measured during polysomnography
Urinary melatonin concentration | At inclusion and at 24 months
  Fractional diuresis
Internal temperature | At inclusion and at 24 months
  The internal temperature will be measured with an e-Celsius capsule during polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Karim BENNYS, MD, Principal Investigator — University Hospital, Montpellier
Locations (3):
- France (3):
  - University Hospital, Montpellier, Montpellier
  - University Hospital of Poitiers, Poitiers
  - University Hospital of Toulouse, Toulouse